CLINICAL TRIAL: NCT05960734
Title: Artificial Intelligence in Healthcare: Advanced Evaluation of Medical Online Content. Assessment of Health Knowledge and Related Educational Intervention.
Brief Title: Artificial Intelligence in Healthcare: Advanced Evaluation of Medical Online Content. AI-driven Quality Assessment of YouTube Videos Providing Information on Incontinence After Cancer Surgery.
Acronym: AMRR UOPhD
Status: Completed | Type: Observational
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Alvaro Manuel Rodriguez Rodriguez, PhD, University of Oviedo
Other Study IDs: AMRR UOPhD
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Cancer; Incontinence; Patient Education; Social Networks; Surgery
Keywords: Cancer; Incontinence; Patient Education; Social Networks; Surgery; Youtube
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Samples group: Samples collected regarding the online information about incontinence after cancer surgery.

SUMMARY:
The aim of the study is to analyse the quality of information that patients and relatives of different types of cancer receive through social networks on the subject of incontinence after cancer surgery.

DETAILED DESCRIPTION:
The primary goal of this study is to meticulously analyze and evaluate the overall quality of information that patients and their relatives obtain through social networks. The specific focus of the investigation lies in exploring the subject of incontinence after cancer surgery, encompassing a diverse range of cancer types. By closely examining the information disseminated across various social platforms, the researchers aim to shed light on the accuracy, reliability, and comprehensiveness of the information available. Ultimately, this study seeks to enhance our understanding of the information landscape surrounding post-cancer surgery incontinence, empowering patients and their relatives to make well-informed decisions regarding their healthcare.

ELIGIBILITY:
Inclusion Criteria:

* Anyone providing information about incontinence after cancer surgery.
* English language

Exclusion Criteria:

* Non-english language
* Duplicated
* Related with advertisements
* Nonrelated to incontinence

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 160 samples providing information about incontinence after cancer surgery.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Analisys of the information in social networks about incontinence after cancer surgery | 2023-2024
  Analisys of the information in social networks about incontinence after cancer surgery

CONTACTS AND LOCATIONS:
Overall Officials: Maria Blanco-Diaz, Prof. PhD., Study Director — University of Oviedo
Locations (1):
- University of Oviedo, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be shared once the study has been completed in its entirety and always respecting the requirements of the Personal Data Protection Law.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 2024-2025
Access Criteria: Via email with the Principal Researcher.